CLINICAL TRIAL: NCT03725059
Title: A Randomized, Double-Blind, Phase III Study of Pembrolizumab Versus Placebo in Combination With Neoadjuvant Chemotherapy and Adjuvant Endocrine Therapy for the Treatment of High-Risk Early-Stage Estrogen Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative (ER+/HER2-) Breast Cancer (KEYNOTE-756)
Brief Title: Study of Pembrolizumab (MK-3475) Versus Placebo in Combination With Neoadjuvant Chemotherapy & Adjuvant Endocrine Therapy in the Treatment of Early-Stage Estrogen Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative (ER+/HER2-) Breast Cancer (MK-3475-756/KEYNOTE-756)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3475-756; MK-3475-756 (Other: MSD); 194604 (Registry Identifier: Japic-CTI); KEYNOTE-756 (Other: MSD); 2023-506921-12-00 (Registry Identifier: EU CT); jRCT2080224535 (Other: jRCT); U1111-1294-6352 (Registry Identifier: UTN); 2017-004869-27 (EudraCT Number)
Record Dates: First submitted 2018-10-29; First posted 2018-10-30 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: PD1; PD-1; PDL1; PD-L1
MeSH Terms: conditions — Breast Neoplasms | interventions — pembrolizumab; Paclitaxel; Doxorubicin; Epirubicin; Cyclophosphamide; Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab+Chemotherapy (KX/KA[E]C) (Experimental): In the neoadjuvant setting, participants receive pembrolizumab (K) 200 mg via intravenous (IV) infusion once every 3 weeks (Q3W) + paclitaxel (X) 80 mg/m^2 via IV infusion once weekly (QW) for 4 cycles (Treatment 1), followed by pembrolizumab 200 mg via IV infusion + doxorubicin or epirubicin (A or E; 60 mg/m^2 or 100 mg/m^2) via IV infusion either in Q2W or Q3W + cyclophosphamide (C) 600 mg/m^2 via IV infusion either in Q2W or Q3W for 4 cycles (Treatment 2). At no more than 6 weeks after last cycle of neoadjuvant treatment, participants will undergo surgery for their breast cancer. After surgery, participants will begin adjuvant study treatment. In the adjuvant setting, participants receive pembrolizumab 200 mg via IV infusion Q3W for 9 cycles + variable endocrine therapy for up to 10 years. Each cycle is 21 days long.
  Interventions: Biological: Pembrolizumab (K); Drug: Paclitaxel (X); Drug: Doxorubicin (A); Drug: Epirubicin (E); Drug: Cyclophosphamide (C); Drug: Endocrine therapy; Radiation: Radiation therapy; Procedure: Surgery
- Placebo+Chemotherapy (PX/PA[E]C) (Placebo Comparator): In the neoadjuvant setting, participants receive placebo (P; normal saline or dextrose) via IV infusion Q3W + paclitaxel (X) 80 mg/m^2 via IV infusion once weekly (QW) for 4 cycles (Treatment 1), followed by placebo via IV infusion + doxorubicin or epirubicin (A or E; 60 mg/m^2 or 100 mg/m^2) via IV infusion either in Q2W or Q3W + cyclophosphamide (C) 600 mg/m^2 via IV infusion either in Q2W or Q3W for 4 cycles (Treatment 2). At no more than 6 weeks after last cycle of neoadjuvant treatment, participants will undergo surgery for their breast cancer. After surgery, participants will begin adjuvant study treatment. In the adjuvant setting, participants receive placebo via IV infusion Q3W for 9 cycles + variable endocrine therapy for up to 10 years. Each cycle is 21 days long.
  Interventions: Drug: Placebo (P); Drug: Paclitaxel (X); Drug: Doxorubicin (A); Drug: Epirubicin (E); Drug: Cyclophosphamide (C); Radiation: Radiation therapy; Procedure: Surgery

INTERVENTIONS:
Biological: Pembrolizumab (K) — IV infusion Q3W
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab+Chemotherapy (KX/KA[E]C)
Drug: Placebo (P) — Normal saline or dextrose IV infusion Q3W
  Arms: Placebo+Chemotherapy (PX/PA[E]C)
Drug: Paclitaxel (X) — IV infusion QW
  Other Names: TAXOL®
Drug: Doxorubicin (A) — IV infusion either in Q2W or Q3W
  Other Names: ADRIAMYCIN®
Drug: Epirubicin (E) — IV infusion either in Q2W or Q3W
  Other Names: ELLENCE®
Drug: Cyclophosphamide (C) — IV infusion either in Q2W or Q3W
  Other Names: CYTOXAN®
Drug: Endocrine therapy — Variable endocrine therapy for up 10 years
  Arms: Pembrolizumab+Chemotherapy (KX/KA[E]C)
Radiation: Radiation therapy — Variable radiation therapy per local standard of care
Procedure: Surgery — Surgery for breast cancer

SUMMARY:
The purpose of this study is to assess the efficacy and safety of pembrolizumab (MK-3475) versus placebo in combination with neoadjuvant (pre-surgery) chemotherapy and adjuvant (post-surgery) endocrine therapy in the treatment of adults who have high-risk early-stage estrogen receptor-positive, human epidermal growth factor receptor 2-negative (ER+/HER2-) breast cancer.

The primary study hypotheses are: 1) pembrolizumab is superior to placebo, both in combination with the protocol-specified neoadjuvant anticancer therapy, as assessed by pathological Complete Response (pCR) rate defined by the local pathologist, and 2) pembrolizumab is superior to placebo (both in combination with the protocol-specified neoadjuvant and adjuvant anticancer therapies) as assessed by Event-Free Survival (EFS) as determined by the investigator. The study is considered to have met its primary objective if pembrolizumab is superior to placebo with respect to either pCR (ypT0/Tis ypN0) or EFS.

DETAILED DESCRIPTION:
Study participants will receive 8 cycles of neoadjuvant study treatment and then will undergo surgery for their breast cancer. After surgery, participants will receive 9 cycles of study treatment and up to 10 years of variable endocrine therapy. Each cycle is 21 days long.

ELIGIBILITY:
Inclusion Criteria:

* Has a localized invasive breast ductal adenocarcinoma, confirmed by the local pathologist, that includes either T1c-T2 (tumor size ≥2 cm), clinical node stage (cN)1-cN2, or T3-T4, cN0-cN2. Note: Inflammatory breast cancer is allowed.
* Has centrally confirmed ER+/HER2-, Grade 3 breast cancer of ductal histology, according to the most recent American Society of Clinical Oncology/College of American Pathologist guidelines.
* Provides a new or recently obtained core needle biopsy, consisting of multiple cores, taken from the primary breast tumor(s) for central determination of HR status (ER and progesterone receptor), HER2, grade, and PD-L1 status.

Note: Sponsor agreement is required for formalin-fixed paraffin-embedded (FFPE) tumor tissue sample or slides that were obtained greater than 60 days prior to the date that the documented informed consent was obtained.

* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, as assessed within 10 days prior to initiation of study treatment.
* Male participants must agree to use contraception during the treatment period and for at least 12 months (for participants who received cyclophosphamide) or 6 months (for participants who did not receive cyclophosphamide) after the last dose of study treatment and refrain from donating sperm during this period.
* Female participants must agree to use effective contraception during the treatment period and for at least 12 months (for participants who received cyclophosphamide) or 6 months (for participants who did not receive cyclophosphamide) after the last dose of study treatment with pembrolizumab or placebo.
* Has adequate organ function.

Exclusion Criteria:

* Has a history of non-infectious pneumonitis that required treatment with steroids or has current pneumonitis.
* Has breast cancer with lobular histology.
* Has bilateral invasive breast cancer.
* Has metastatic (Stage IV) breast cancer.
* Has multi-centric breast cancer (presence of more than 1 tumor in different quadrants of the breast).
* Has any of the following clinical lymph node staging per current American Joint Committee on Cancer (AJCC) staging criteria for breast cancer staging based on radiological and/or clinical assessment: cN3, cN3a, cN3b, or cN3c.
* Has ER-, progesterone receptor positive breast cancer.
* Has undergone excisional biopsy of the primary tumor and/or axillary lymph nodes or has undergone sentinel lymph node biopsy prior to study treatment.
* Has a known additional, invasive, malignancy that is progressing or required active treatment in the last 5 years.

Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, ductal breast carcinoma in situ, or cervical carcinoma in situ that has undergone potentially curative therapy are not excluded.

* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs) Note: Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
* Has a known history of active tuberculosis (Bacillus tuberculosis).
* Has an active infection requiring systemic therapy.
* Has left ventricular ejection fraction (LVEF) of <50% or below the institution limit of normal, as assessed by echocardiogram (ECHO) or multigated acquisition (MUGA) scan performed at screening.
* Has other significant cardiac disease, such as: 1) History of myocardial infarction, acute coronary syndrome, or coronary angioplasty/stenting/bypass within the last 6 months. or 2) Congestive heart failure (CHF) New York Heart Association (NYHA) Class II-IV or history of CHF NYHA Class III or IV.
* Has a known history of human immunodeficiency virus (HIV) infection.
* Has a known history of hepatitis B or known active hepatitis C virus infection.
* Has received prior treatment for breast cancer.
* Has received prior therapy with an anti-programmed cell death protein 1 (anti-PD-1), anti-programmed cell death-ligand 1 (anti-PD-L1), or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g. cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], OX 40, CD137).
* Has received a live vaccine within 30 days prior to the first dose of study treatment.
* Has severe hypersensitivity (≥Grade 3) to any of the components or excipients used in the study treatments.
* Is/was enrolled in a study of an investigational agent and received study therapy, or used an investigational device within 4 weeks (12 months for an investigational agent or device with anticancer or antiproliferative properties) prior to the first dose of study treatment.
* Is pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 12 months (for participants who received cyclophosphamide) or 6 months (for participants who did not receive cyclophosphamide) after the last dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1240 (Estimated)
Dates: Start 2018-12-27 (Actual); Primary Completion 2031-01-24 (Estimated); Study Completion 2031-01-24 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) Rate Using the Definition of ypT0/Tis ypN0 | Up to approximately 7 months (Time of surgery)
  The pCR rate (ypT0/Tis ypN0) is defined as the percentage of participants without residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy by American Joint Committee on Cancer (AJCC) staging criteria (8th edition) assessed by the local pathologist at the time of surgery. The percentage of participants with a pathological Complete Response (pCR) using the definition of (ypT0/Tis ypN0) will be presented for pembrolizumab versus placebo, both in combination with the protocol-specified neoadjuvant anticancer therapies.
Event-Free Survival (EFS) | Up to approximately 12 years
  EFS is defined as the time from randomization to disease progression that: precludes surgery, results in a local or distant recurrence, results in a second primary malignancy, or death due to any cause whichever occurs first. The EFS following administration of pembrolizumab and placebo, both in combination with the protocol-specified neoadjuvant and adjuvant anticancer therapies, as determined by the investigator will be presented.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 12 years
  OS is defined as the time from date of randomization to date of death due to any cause. The OS following administration of pembrolizumab and placebo, both in combination with the protocol-specified neoadjuvant and adjuvant anticancer therapies will be presented.
pCR Rate Using the Definition of ypT0ypN0 | Up to approximately 7 months (Time of surgery)
  pCR rate (ypT0ypN0) is defined as the percentage of participants without residual invasive or in situ cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes after completion of neoadjuvant systemic therapy by AJCC staging criteria (8th edition) assessed by the local pathologist at the time of surgery. The percentage of participants with a pCR using the definition of (ypT0ypN0) will be presented for pembrolizumab versus placebo, both in combination with the protocol-specified neoadjuvant anticancer therapies.
pCR Rate Using the Definition of ypT0/Tis | Up to approximately 7 months (Time of surgery)
  pCR rate (ypT0/Tis) is defined as the percentage of participants without residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen (independent of lymph node involvement) after completion of neoadjuvant systemic therapy by AJCC staging criteria (8th edition) assessed by the local pathologist at the time of surgery. The percentage of participants with a pCR using the definition of ypT0/Tis will be presented for pembrolizumab versus placebo, both in combination with the protocol-specified neoadjuvant anticancer therapies.
pCR Rate Using the Definitions of ypT0/Tis ypN0, ypT0/Tis, and ypT0 ypN0 in Participants With a Combined Positive Score [CPS] ≥1 | Up to approximately 7 months (Time of surgery)
  pCR rates were calculated using the definitions of ypT0/Tis ypN0, ypT0/Tis, and ypT0 ypN0 after completion of neoadjuvant systemic therapy by AJCC staging criteria (8th edition) assessed by the local pathologist at the time of surgery. The percentage of participants with a pCR using the three definitions of ypT0/Tis ypN0, ypT0/Tis, and ypT0 ypN0 in participants with a CPS ≥1 (with a positive Programmed Cell Death-Ligand 1 [PD-L1] tumor status) will be presented for pembrolizumab versus placebo, both in combination with the protocol-specified neoadjuvant anticancer therapies.
EFS in Participants With a CPS ≥1 | Up to approximately 12 years
  EFS is defined as the time from randomization to disease progression that: precludes surgery, results in a local or distant recurrence, results in a second primary malignancy, or death due to any cause whichever occurs first. The EFS following administration of pembrolizumab and placebo, both in combination with the protocol-specified neoadjuvant and adjuvant anticancer therapies, as determined by the investigator for participants with a CPS ≥1 will be presented.
OS in Participants With a CPS ≥1 | Up to approximately 12 years
  OS is defined as the time from date of randomization to date of death due to any cause. The OS following administration of pembrolizumab and placebo, both in combination with the protocol-specified neoadjuvant and adjuvant anticancer therapies for participants with a CPS ≥1 will be presented.
Number of Participants Experiencing an Adverse Event (AE) | Up to approximately 15 months
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience an AE while receiving pembrolizumab or placebo (including 1 month of safety follow up) will be presented.
Number of Participants Experiencing a Serious Adverse Event (SAE) | Up to approximately 17 months
  An SAE is defined as any untoward medical occurrence that, at any dose: Results in death, Is life-threatening, Requires inpatient hospitalization or prolongation of existing hospitalization, Results in persistent or significant disability/incapacity or Is a congenital anomaly/birth defect. The number of participants who experience an SAE while receiving pembrolizumab or placebo (including 3 months of safety follow up) will be presented.
Number of Participants Experiencing an Immune-related AE (irAE) | Up to approximately 15 months
  Some AEs that may occur in this study that are known to be related to pembrolizumab immunotherapy treatment and may include: pneumonitis, diarrhea/colitis, aspartate aminotransferase/alanine aminotransferase (AST/ALT) elevation or increased bilirubin, Type 1 diabetes mellitus or hyperglycemia, hypophysitis, hyperthyroidism, hypothyroidism, nephritis and renal dysfunction, and myocarditis. The number of participants who experience an irAE while receiving pembrolizumab or placebo (including 1 month of safety follow up) will be presented.
Number of Participants who Discontinued Study Treatment Due to an AE | Up to approximately 14 months
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinue study treatment (pembrolizumab or placebo) due to an AE will be presented.
Change from Baseline in European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life (QoL) Questionnaire Core 30 (QLQ-C30) Score | Baseline (Cycle 1 Day 1 in Treatment 1) and Cycles 1 and 4 Day 1 in Treatment 2 (Up to approximately 5 months) Each cycle is 21 days.
  The EORTC QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Individual responses for each of 28 items are given on a 4-point scale (1=Not at All to 4=Very Much), with a lower score indicating a better outcome, and responses for each of 2 items (overall health and overall quality of life) are given on a 7-point scale (1=Very poor to 7=Excellent), with a higher score indicating a better outcome. The change from Baseline to end of treatment (up to Cycle 4 Day 1) in EORTC-QLQ-C30 scores for participants will be presented.
Change from Baseline in EORTC Breast Cancer-Specific QoL Questionnaire (QLQ-BR23) Score | Baseline (Cycle 1 Day 1 in Treatment 1) and Cycles 1 and 4 Day 1 in Treatment 2 (Up to approximately 5 months) Each cycle is 21 days.
  The EORTC QLQ-BR23 is a 23-item questionnaire developed to assess the quality of life in women with breast cancer. Responses for each item are given on a 4-point scale (1=Not at All to 4=Very Much), with a lower score indicating a better outcome. The change from Baseline to end of treatment (up to Cycle 4 Day 1) in EORTC QLQ-BR23 score for participants will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (244):
- United States (45):
  - Southern Cancer Center, PC ( Site 8003), Daphne, Alabama
  - Cancer Treatment Centers of America at Western Regional Medical Center ( Site 0001), Goodyear, Arizona
  - Arizona Oncology Associates PC- HOPE ( Site 8008), Tucson, Arizona
  - Cedars Sinai Medical Center Samuel Oschin Comp. Cancer Institute ( Site 0079), Los Angeles, California
  - El Camino Hospital Cancer Center ( Site 0004), Mountain View, California
  - Stanford Cancer Center ( Site 0072), Palo Alto, California
  - UC Davis Comprehensive Cancer Center ( Site 0073), Sacramento, California
  - University of Colorado, Anschutz Cancer Pavilion ( Site 0008), Aurora, Colorado
  - Baptist MD Anderson Cancer Center ( Site 0014), Jacksonville, Florida
  - Southeastern Regional Medical Center, Inc. ( Site 0075), Newnan, Georgia
  - The University of Chicago Medical Center ( Site 0080), Chicago, Illinois
  - Orchard Healthcare Research Inc. ( Site 0020), Skokie, Illinois
  - Midwestern Regional Medical Center, Inc. ( Site 0077), Zion, Illinois
  - Goshen Center for Cancer Care ( Site 0021), Goshen, Indiana
  - MercyOne Waterloo Cancer Center ( Site 0016), Waterloo, Iowa
  - James Graham Brown Cancer Center ( Site 0022), Louisville, Kentucky
  - Maryland Oncology Hematology, P.A. ( Site 8007), Bethesda, Maryland
  - Massachusetts General Hospital ( Site 0024), Boston, Massachusetts
  - MGH - North Shore Cancer Center ( Site 0081), Danvers, Massachusetts
  - MGH Newton-Wellesley Hospital's Vernon Cancer Center ( Site 0082), Newton, Massachusetts
  - Henry Ford Health System ( Site 0028), Detroit, Michigan
  - Mayo Clinic and Medical School (Rochester) ( Site 0029), Rochester, Minnesota
  - St. Vincent Frontier Cancer Center ( Site 0033), Billings, Montana
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists ( Site 0039), Omaha, Nebraska
  - Holy Name Medical Center ( Site 0041), Teaneck, New Jersey
  - Weill Cornell Medical College ( Site 0043), New York, New York
  - CTCA Southwestern ( Site 0074), Tulsa, Oklahoma
  - OHSU Knight Cancer Institute ( Site 0051), Portland, Oregon
  - Northwest Cancer Specialists, P.C. ( Site 8000), Tigard, Oregon
  - Geisinger Medical Center ( Site 0052), Danville, Pennsylvania
  - Fox Chase Cancer Center ( Site 0078), Philadelphia, Pennsylvania
  - Cancer Treatment Centers of America-Eastern Regional Medical Center ( Site 0076), Philadelphia, Pennsylvania
  - Medical University of South Carolina ( Site 0053), Charleston, South Carolina
  - Tennessee Oncology, PLLC/The Sarah Cannon Research Institute ( Site 7000), Nashville, Tennessee
  - Texas Oncology-Austin Central ( Site 8004), Austin, Texas
  - Texas Oncology-Dallas Presbyterian Hospital ( Site 8002), Dallas, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center ( Site 8009), Dallas, Texas
  - Texas Oncology-Memorial City ( Site 8012), Houston, Texas
  - University of Texas-MD Anderson Cancer Center ( Site 0083), Houston, Texas
  - Texas Oncology- Plano East ( Site 8010), Plano, Texas
  - Texas Oncology - Northeast Texas ( Site 8006), Tyler, Texas
  - Bon Secours St. Francis Medical Center Oncology Research ( Site 0064), Midlothian, Virginia
  - Virginia Oncology Associates ( Site 8001), Norfolk, Virginia
  - Kadlec Clinic Hematology and Oncology ( Site 0070), Kennewick, Washington
  - Medical Oncology Associates (Summit Cancer Centers) ( Site 0066), Spokane, Washington
- Australia (6):
  - Chris OBrien Lifehouse ( Site 2107), Camperdown, New South Wales
  - Royal North Shore Hospital ( Site 2100), Sydney, New South Wales
  - Westmead Hospital ( Site 2101), Sydney, New South Wales
  - Mater Misericordiae Ltd ( Site 2106), South Brisbane, Queensland
  - Frankston Hospital ( Site 2103), Frankston, Victoria
  - Peter MacCallum Cancer Centre ( Site 2102), Melbourne, Victoria
- Belgium (10):
  - Imelda Ziekenhuis Bonheiden ( Site 0703), Bonheiden, Antwerpen
  - UZ Antwerpen - Medical Oncology ( Site 0709), Edegem, Antwerpen
  - Institut Jules Bordet ( Site 0710), Anderlecht, Bruxelles-Capitale, Region de
  - Cliniques Universitaires Saint-Luc ( Site 0701), Brussels, Bruxelles-Capitale, Region de
  - CHC MontLegia ( Site 0707), Liège, Liege
  - Jessa Ziekenhuis Campus Virga Jesse ( Site 0704), Hasselt, Limburg
  - CHU UCL Namur Site de Godinne ( Site 0706), Yvoir, Namur
  - AZ Maria Middelares Gent ( Site 0700), Ghent, Oost-Vlaanderen
  - UZ Leuven ( Site 0702), Leuven, Vlaams-Brabant
  - AZ Groeninge ( Site 0705), Kortrijk, West-Vlaanderen
- Brazil (10):
  - Hospital Araujo Jorge Associacao de Combate ao Cancer de Goias ( Site 0205), Goiânia, Goiás
  - ONCOSITE - Centro de Pesquisa Clinica em Oncologia ( Site 0206), Ijuí, Rio Grande do Sul
  - Associacao Hospitalar Moinhos de Vento ( Site 0201), Porto Alegre, Rio Grande do Sul
  - Uniao Brasileira de Educacao e Assistencia Hospital Sao Lucas da Pucrs ( Site 0202), Porto Alegre, Rio Grande do Sul
  - CEPON - Centro de Pesquisas Oncologicas ( Site 0208), Florianópolis, Santa Catarina
  - Centro de Novos Tratamentos Itajai - Clinica de Neoplasias Litoral ( Site 0207), Itajaí, Santa Catarina
  - Instituto Nacional de Câncer - INCA-Pesquisa Clinica HC3 ( Site 0200), Rio de Janeiro
  - Clinica de Pesquisas e Ctro de Estudos Onc. Ginecol. e Mamaria Ltda ( Site 0204), São Paulo
  - Núcleo de Pesquisa Clínica da Rede São Camilo ( Site 0210), São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP ( Site 0209), São Paulo
- Canada (9):
  - Cross Cancer Institute ( Site 0115), Edmonton, Alberta
  - BC Cancer-Vancouver Center ( Site 0116), Vancouver, British Columbia
  - Princess Margaret Cancer Centre ( Site 0112), Toronto, Ontario
  - CISSS de la Monteregie-Centre ( Site 0108), Greenfield Park, Quebec
  - Hopital Maisonneuve-Rosemont CIUSSS de l Est de L Ile de Montreal ( Site 0111), Montreal, Quebec
  - Centre Hospitalier de l Universite de Montreal - CHUM ( Site 0114), Montreal, Quebec
  - Jewish General Hospital ( Site 0103), Montreal, Quebec
  - CHU de Quebec Universite Laval - Hopital du Saint-Sacrement ( Site 0101), Québec, Quebec
  - Centre Hospitalier Regional de Trois-Rivieres ( Site 0106), Trois-Rivières, Quebec
- China (18):
  - Anhui Provincial Hospital ( Site 3224), Heifei, Anhui
  - Ruijin Hosp,Shanghai Jiao Tong University School of Medicine ( Site 3215), Shanghai, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences ( Site 3208), Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital-1 Bingfanglou-Oncology ( Site 3207), Fuzhou Fujian, Fujian
  - Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University ( Site 3213), Guangzhou, Guangdong
  - Fourth Hospital Of Hebei Medical University ( Site 3216), Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital ( Site 3200), Harbin, Heilongjiang
  - Henan Cancer Hospital ( Site 3212), Zhengzhou, Henan
  - Hubei Cancer Hospital ( Site 3211), Wuhan, Hubei
  - Hunan Cancer Hospital ( Site 3214), Changsha, Hunan
  - The First Affiliated Hospital of Zhejiang University ( Site 3203), Hangzhou, Jiangsu
  - The First Hospital of Jilin University ( Site 3201), Changchun, Jilin
  - Fudan University Shanghai Cancer Center ( Site 3205), Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi an Jiaotong University ( Site 3220), Xi’an, Shanxi
  - Tianjin Medical University Cancer Institute & Hospital ( Site 3209), Tianjin, Tianjin Municipality
  - The Affiliated Cancer Hospital of Xinjiang Medical ( Site 3219), Ürümqi, Xinjiang
  - Zhejiang Provincial People's Hospital ( Site 3225), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital ( Site 3210), Hangzhou, Zhejiang
- Colombia (7):
  - Fundacion Colombiana de Cancerología Clinica Vida ( Site 0405), Medellín, Antioquia
  - Rodrigo Botero SAS ( Site 0407), Medellín, Antioquia
  - Clinica de la Costa S.A.S. ( Site 0400), Barranquilla, Atlántico
  - Centro de Investigacion Clinica del Country ( Site 0402), Bogotá, Bogota D.C.
  - Fundacion Universitaria Sanitas ( Site 0403), Bogotá, Bogota D.C.
  - IMAT S.A.S ( Site 0401), Montería, Departamento de Córdoba
  - Clínica Imbanaco S.A.S ( Site 0406), Cali, Valle del Cauca Department
- Hospital Metropolitano - Sede Lindora ( Site 4203), Santa Ana, Provincia de San José, Costa Rica
- France (14):
  - Centre Francois Baclesse ( Site 0927), Caen, Calvados
  - Centre Georges Francois Leclerc ( Site 0920), Dijon, Cote-d Or
  - Institut Claudius Regaud IUCT Oncopole ( Site 0903), Toulouse, Haute-Garonne
  - Centre Oscar Lambret ( Site 0911), Lille, Hauts-de-France
  - Institut Curie - Centre Rene Huguenin ( Site 0917), Saint-Cloud, Hauts-de-Seine
  - Centre de Cancerologie du Grand Montpellier ( Site 0925), Montpellier, Herault
  - CHR-METZ-THIONVILLE - Hopital de Mercy ( Site 0919), Metz, Moselle
  - Institut Sainte Catherine ( Site 0916), Avignon, Provence-Alpes-Côte d'Azur Region
  - Centre Jean Perrin ( Site 0909), Clermont-Ferrand, Puy-de-Dome
  - Clinique Victor Hugo Le Mans ( Site 0906), Le Mans, Sarthe
  - Institut Gustave Roussy ( Site 0926), Villejuif, Val-de-Marne
  - Institut Curie ( Site 0900), Paris
  - Hopital Saint-Louis ( Site 0908), Paris
  - Hopital Tenon ( Site 0914), Paris
- Germany (12):
  - Medizinische Management GmbH ( Site 1012), Friedrichshafen, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen ( Site 1001), Erlangen, Bavaria
  - Klinikum der Universitaet Muenchen - Grosshadern ( Site 1000), Munich, Bavaria
  - Sana Klinikum Offenbach GmbH ( Site 1002), Offenbach, Hesse
  - HELIOS Dr. Horst Schmidt Kliniken Wiesbaden ( Site 1004), Wiesbaden, Hesse
  - MVZ Onko Medical GmbH Hannover ( Site 1013), Hanover, Lower Saxony
  - Gynaekologisches Zentrum ( Site 1003), Bonn, North Rhine-Westphalia
  - Kliniken Essen Mitte Gmbh Evang. Huyssens Stiftung ( Site 1006), Essen, North Rhine-Westphalia
  - Frauenklinik St. Louise ( Site 1014), Paderborn, North Rhine-Westphalia
  - Caritas Klinikum Saarbruecken St. Theresia ( Site 1009), Saarbrücken, Saarland
  - Universitaetsklinikum Carl Gustav Carus ( Site 1008), Dresden, Saxony
  - MVZ Nordhausen gGmbH - Praxis Dr. Grafe ( Site 1005), Nordhausen, Thuringia
- Hungary (8):
  - Pecsi Tudomanyegyetem Klinikai Kozpont ( Site 2905), Pécs, Baranya
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi OktatoKorhaz ( Site 2904), Miskolc, Borsod-Abauj Zemplen county
  - Bacs-Kiskun Varmegyei Oktatokorhaz-Onkoradiologiai Kozpont ( Site 2913), Kecskemét, Bács-Kiskun county
  - Budapesti Szent Margit Korhaz ( Site 2901), Budapest
  - Orszagos Onkologiai Intezet ( Site 2908), Budapest
  - Budapesti Uzsoki Utcai Kórház-Onkoradiológiai Osztály ( Site 2902), Budapest
  - Debreceni Egyetem Klinikai Kozpont ( Site 2907), Debrecen
  - Somogy Megyei Kaposi Mor Oktato Korhaz ( Site 2915), Kaposvár
- Ireland (2):
  - Bon Secours Hospital ( Site 1554), Cork
  - St. James s Hospital ( Site 1553), Dublin
- Israel (13):
  - HaEmek Medical Center ( Site 1712), Afula
  - Assuta Ashdod Public ( Site 1704), Ashdod
  - Soroka Medical Center ( Site 1701), Beersheba
  - Rambam Health Care Campus-Oncology Division ( Site 1705), Haifa
  - Shaare Zedek Medical Center ( Site 1708), Jerusalem
  - Hadassah Ein Karem - Sharett Institute of Oncology ( Site 1700), Jerusalem
  - Meir Medical Center ( Site 1710), Kfar Saba
  - Holy Family Hospital ( Site 1711), Nazareth
  - Rabin Medical Center ( Site 1702), Petah Tikva
  - Chaim Sheba Medical Center. ( Site 1707), Ramat Gan
  - Kaplan Medical Center ( Site 1703), Rehovot
  - Sourasky Medical Center ( Site 1706), Tel Aviv
  - Assuta Medical Center ( Site 1709), Tel Aviv
- Japan (16):
  - Aichi Cancer Center ( Site 2601), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 2613), Kashiwa, Chiba
  - National Hospital Organization Hokkaido Cancer Center ( Site 2607), Sapporo, Hokkaido
  - Hyogo Medical University Hospital ( Site 2600), Nishinomiya, Hyōgo
  - Kitasato University Hospital ( Site 2616), Sagamihara, Kanagawa
  - Kumamoto University Hospital ( Site 2602), Kumamoto, Kumamoto
  - Saitama Medical University International Medical Center ( Site 2606), Hidaka, Saitama
  - Saitama Prefectural Cancer Center ( Site 2612), Kitaadachi-gun, Saitama
  - Shizuoka Cancer Center ( Site 2611), Suntogun, Shizuoka
  - Chiba Cancer Center ( Site 2605), Chiba
  - Fukushima Medical University Hospital ( Site 2610), Fukushima
  - Hiroshima City Hiroshima Citizens Hospital ( Site 2603), Hiroshima
  - National Hospital Organization Osaka National Hospital ( Site 2614), Osaka
  - Toranomon Hospital ( Site 2608), Tokyo
  - Cancer Institute Hospital of JFCR ( Site 2604), Tokyo
  - Showa Medical University Hospital ( Site 2615), Tokyo
- New Zealand (3):
  - Tauranga Hospital ( Site 2302), Tauranga, Bay of Plenty
  - Canterbury Regional Cancer & Blood Services ( Site 2303), Christchurch, Canterbury
  - Capital & Coast District Health Board - Wellington Hospital ( Site 2301), Wellington
- Poland (12):
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka ( Site 1800), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Dolnoslaskie Centrum Onkologii. ( Site 1820), Wroclaw, Lower Silesian Voivodeship
  - Mazowiecki Szpital Specjalistyczny im. dr Jozefa Psarskiego ( Site 1814), Ostrołęka, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie ( Site 1899), Warsaw, Masovian Voivodeship
  - Mazowiecki Szpital Onkologiczny ( Site 1803), Wieliszew, Masovian Voivodeship
  - Bialostockie Centrum Onkologii ( Site 1819), Bialystok, Podlaskie Voivodeship
  - Wojewodzkie Centrum Onkologii Copernicus ( Site 1817), Gdansk, Pomeranian Voivodeship
  - Szpitale Pomorskie Sp. z o.o. ( Site 1818), Gdynia, Pomeranian Voivodeship
  - Beskidzkie Centrum Onkologii im. Jana Pawla II ( Site 1810), Bielsko-Biala, Silesian Voivodeship
  - Wojewodzki Szpital Specjalistyczny nr 4 w Bytomiu ( Site 1807), Bytom, Silesian Voivodeship
  - Narodowy Instytut Onkologii - Oddzial w Gliwicach ( Site 1801), Gliwice, Silesian Voivodeship
  - Instytut Centrum Zdrowia Matki Polki ( Site 1821), Lodz, Łódź Voivodeship
- Portugal (4):
  - Fundacao Champalimaud ( Site 2500), Lisboa, Aveiro District
  - Unidade Local de Saude de Santa Maria - Hospital de Santa Maria ( Site 2501), Lisbon
  - Unidade Local de Saude de Santo António - Hospital Santo António ( Site 2503), Porto
  - Inst. Portugues de Oncologia de Porto Francisco Gentil EPE ( Site 2502), Porto
- UPR Comprehensive Cancer Center ( Site 6200), San Juan, Puerto Rico
- Russia (10):
  - Arkhangelsk Clinical Oncological Dispensary ( Site 1901), Arkhangelsk, Arkhangelskaya oblast
  - Republican Clinical Oncology Dispensary of Republic of Bashkortostan ( Site 1909), Ufa, Baskortostan, Respublika
  - N.N. Blokhin NMRCO ( Site 1908), Moscow, Moscow
  - Central Clinical Hospital with outpatient Clinic ( Site 1907), Moscow, Moscow
  - Medical Rehabilitation Center ( Site 1912), Moscow, Moscow
  - Ryazan Regional Clinical Oncology Dispensary ( Site 1910), Ryazan, Ryazan Oblast
  - Railway Hospital of OJSC ( Site 1913), Saint Petersburg, Sankt-Peterburg
  - Scientific Research Oncology Institute n.a. N.N.Petrov ( Site 1900), Saint Petersburg, Sankt-Peterburg
  - Republican Clinical Oncology Dispensary of Tatarstan MoH named after professor M.Z. Sigal ( Site 1903), Kazan', Tatarstan, Respublika
  - Tomsk Scientific Research Institute of Oncology ( Site 1905), Tomsk, Tomsk Oblast
- South Korea (5):
  - National Cancer Center ( Site 2204), Goyang-si, Kyonggi-do
  - Seoul National University Hospital ( Site 2200), Seoul
  - Severance Hospital Yonsei University Health System ( Site 2201), Seoul
  - Asan Medical Center ( Site 2202), Seoul
  - Samsung Medical Center ( Site 2203), Seoul
- Spain (14):
  - Instituto Catalan de Oncologia ICO - Hospital Duran i Reynals ( Site 1363), L'Hospitalet de Llobregat, Barcelona
  - Hospital Teresa Herrera - Chuac ( Site 1358), A Coruña, La Coruna
  - Hospital Quiron de Madrid ( Site 1351), Pozuelo de Alarcón, Madrid
  - Hospital General Universitario Gregorio Maranon ( Site 1367), Madrid, Madrid, Comunidad de
  - Hospital Clinico Universitario de Valencia ( Site 1355), Valencia, Valenciana, Comunitat
  - Instituto Oncologico Baselga.Hospital Quiron. ( Site 1352), Barcelona
  - Hospital Vall D Hebron ( Site 1357), Barcelona
  - Hospital Clinic I Provincial de Barcelona ( Site 1353), Barcelona
  - Complejo Hospitalario de Jaen ( Site 1364), Jaén
  - Hospital Beata María Ana-oncology ( Site 1370), Madrid
  - Hospital Clinico San Carlos ( Site 1354), Madrid
  - Hospital Universitario 12 de Octubre ( Site 1356), Madrid
  - Hospital Universitario Virgen del Rocio ( Site 1360), Seville
  - Hospital General Arnau de Vilanova de Valencia ( Site 1369), Valencia
- Taiwan (5):
  - China Medical University Hospital ( Site 2401), Taichung
  - National Cheng Kung University Hospital ( Site 2400), Tainan
  - National Taiwan University Hospital ( Site 2404), Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center ( Site 2403), Taipei
  - Linkou Chang Gung Memorial Hospital ( Site 2402), Taoyuan District
- Ukraine (11):
  - MNPE City Clinical Hospital #4 of Dnipro Regional Council ( Site 2702), Dnipro, Dnipropetrovsk Oblast
  - MI Kryviy Rih Center of Dnipropetrovsk Regional Council ( Site 2700), Kryviy Rih, Dnipropetrovsk Oblast
  - MI Precarpathian Clinical Oncology Center ( Site 2707), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Communal non profit enterprise Regional Clinical Oncology Center ( Site 2721), Kharkiv, Kharkivs’ka Oblast’
  - Communal nonprofit enterprise "Kherson Regional Oncology Dispensary" of Kherson Regional Council ( Site 2713), Antonivka Village, Kherson Oblast
  - Khmelnitskiy Regional Onkology Dispensary ( Site 2704), Khmelnitskiy, Khmelnytskyi Oblast
  - SNPE National Cancer Institute ( Site 2719), Kyiv, Kyivska Oblast
  - MI Odesa Regional Clinical Hospital ( Site 2701), Odesa, Odesa Oblast
  - MI Odessa Regional Oncological Centre ( Site 2714), Odesa, Odesa Oblast
  - Medical center of the Limited Liability Company Yulis ( Site 2720), Zaporizhzhia, Zaporizhzhia Oblast
  - Kyiv City Clinical Oncology Centre ( Site 2716), Kyiv
- United Kingdom (8):
  - University Hospitals Bristol NHS Foundation Trust ( Site 1503), Bristol, Bristol, City of
  - Nottingham University Hospitals NHS Trust ( Site 1504), Nottingham, England
  - Colchester General Hospital ( Site 1508), Colchester, Essex
  - Barts Health NHS Trust ( Site 1500), London, London, City of
  - Guy's Hospital ( Site 1501), London, London, City of
  - St. Georges University Hospital NHS Foundation Trust ( Site 1505), London, London, City of
  - Birmingham & Solihull Heartlands Hospital NHS ( Site 1506), Solihull
  - Royal Cornwall Hospital ( Site 1502), Truro

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Cardoso F, O'Shaughnessy J, Liu Z, McArthur H, Schmid P, Cortes J, Harbeck N, Telli ML, Cescon DW, Fasching PA, Shao Z, Loirat D, Park YH, Fernandez MG, Rubovszky G, Spring L, Im SA, Hui R, Takano T, Andre F, Yasojima H, Ding Y, Jia L, Karantza V, Tryfonidis K, Bardia A. Pembrolizumab and chemotherapy in high-risk, early-stage, ER+/HER2- breast cancer: a randomized phase 3 trial. Nat Med. 2025 Feb;31(2):442-448. doi: 10.1038/s41591-024-03415-7. Epub 2025 Jan 21. PMID 39838117
- [Derived] Schlam I, Corti C, Sammons S, Mittendorf EA, Tolaney SM. Checkpoint inhibition for early-stage hormone receptor-positive breast cancer. Expert Opin Biol Ther. 2024 Jun;24(6):511-520. doi: 10.1080/14712598.2024.2370395. Epub 2024 Jun 24. PMID 38913933
- See also: Merck Clinical Trials Information — https://merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26258&tenant=MT_MSD_9011